CLINICAL TRIAL: NCT06058637
Title: Online Nurse-assisted Eye-screening in Home Healthcare; Implementation Study and Economic Evaluation, From an Individual, Healthcare and Socio-political Perspective
Brief Title: iSCREEN-study: Online Nurse-assisted Eye-screening in Home Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Easee B.V. (Unknown)
Responsible Party: Principal Investigator, R.M.A. (Ruth) van Nispen, Prof.dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NL78386.029.21
Record Dates: First submitted 2023-07-03; First posted 2023-09-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Eye Diseases
Keywords: Eye screening; Elderly; Home healthcare; Visual impairment; Cluster randomized controlled trial
MeSH Terms: conditions — Eye Diseases; Vision Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Research assistants who will perform the measurements after randomisation will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual (No Intervention)
- Eye screening on top of care (Experimental)
  Interventions: Device: Eye screening

INTERVENTIONS:
Device: Eye screening — Nurse-assisted eye-screening will take place with the Easee app, which is implemented on the tablet or laptop of the community nurse. The nurse's smartphone will function as a remote control by which he/she submits input to a computer screen that displays the test. If the participant can do the test by him or herself, the nurse will merely supervise to ensure correct application. Standard audio instructions guide the nurse and participant through the test. The test will start with triage questions, which are used to set up a correct referral. During the test, both eyes are tested consecutively, covering one eye at a time. The participant will wear his/her spectacles, if present. The participant is presented a sequence of optotypes (i.e. tumbling-E and triangle-circle optotypes) that the participant must correctly identify, in addition to various grate sizes, both near and at a distance. The Amsler grid test is performed to detect any macular problems.
  Arms: Eye screening on top of care

SUMMARY:
The aim of this study is to investigate the cost-effectiveness of a nurse-assisted online eye-screening in home healthcare in reducing eye complaints.

DETAILED DESCRIPTION:
Background:

In the Netherlands, the prevalence of blindness and low vision is highest among the elderly in care institutions and in home healthcare (20-25%). A recent cross-sectional pilot study with one of the largest home healthcare organizations in the Netherlands (i.e. 'Buurtzorg Nederland') showed that simple eye-screening by community nurses helps to detect eye complaints among elderly people living independently. Of all patients who were referred to a general practitioner (GP), optician, optometrist or ophthalmologist based on this screening (20% of the total group), it was found that almost half had severe visual impairment, whereas others had eye complaints that had affected acuity to a smaller extent. In most cases, eye complaints could be treated with spectacles or cataract surgery, but also untreatable eye diseases were found. These complaints may not have been detected without eye-screening and treatment would not have been offered. Often, the elderly themselves or family/friends or care providers, do not recognize that their eyesight has decreased. However, this can negatively affect their quality of life and health status. To increase access to eye care the investigators will perform a study using an online eye screening, which can be performed by the community nurses or possibly the participants themselves in their home environment.

Purpose:

The aim of this study is to investigate the cost-effectiveness of a nurse-assisted online eye-screening in home healthcare in reducing eye complaints.

Method:

The investigators will perform a cluster-RCT to compare online eye-screening guided by community nurses in addition to care as usual to a control condition, receiving only care as usual. It will be performed in collaboration with several home healthcare organizations. Measurements in both groups will take place at baseline, after 6 months and 12 months. This will include visual acuity measurements, questionnaires and an optometric examination.

This study will be conducted among 220 participants. Elderly clients, 65+, who receive home healthcare will be invited to participate. Clients who have a serious health condition, clients who are cognitively unable to participate, or clients who had received an optometric consultation within the last 6 months, will be excluded.

The eye-screening is developed by Easee and is CE marked. During the test, the visual acuity will be measured both near and at distance, and the Amsler grid test will be performed. The results of the eye-screening will be checked by an optometrist, and will be made available to the participant. This will be done by letter including a recommendation for a referral, if necessary.

ELIGIBILITY:
Inclusion criteria

* Patients receive home healthcare for health problems
* 65 years or older
* Understanding of the Dutch language
* Cognitive ability to participate in research (six-item Mini Mental State Examination: score >3)

Exclusion criteria

* Very serious health condition of the patient (i.e. terminal illness, receiving palliative home care)
* Cognitively unable to participate in research (e.g. late stage Alzheimer's/Dementia, Parkinson's) (six-item Mini Mental State Examination: score ≤3)
* Having received an optometric or ophthalmic consultation within the last 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 234 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Colenbrander-1M visual acuity | 12 months
  Incidence in clinically relevant change of 2 lines or more on the Colenbrander-1M visual acuity chart

SECONDARY OUTCOMES:
Colenbrander-1M visual acuity change | 12 months
  Average visual acuity change per eye in letters
Colenbrander-1M visual acuity change in participants with baseline visual impairment | 12 months
  Number of participants with baseline visual impairment and clinically relevant change of 2 lines or more on the Colenbrander-1M visual acuity
Optometric status | 12 months
  Optometric status assessed by slitlamp/fundusfotography
Vision related quality of life with the EyeQ questionnaire | 12 months
  EyeQ questionnaire with 46 items. The items can be scored from "never" to always". EyeQ scores are expressed on a theta logit-scale from -4 (highest vision related quality of life) to +4 (lowest vision related quality of life).
Amsler grid chart | 12 months
  The Amsler grid is a simple square containing a grid pattern and a dot in the middle. It is used to detect symptoms of macular degeneration. The chart is held at a distance of 30 cm. Single eye test will be done. A participant is asked to look at the central dot of the Amsler grid chart. In normal cases, the lines of the chart will be seen straight and parallel. 4 questions will be used to notice abnormalities such as distortion of lines, broken lines, missing lines and wavy lines.
Fall and fracture calendar | 12 months
  Falling accidents and bone fractures will be assessed with a shortened version of the 'fall and fracture calendar'. A questionnaire with 6 questions on the number of falls and fractures during the last 6 months.
Depressive symptomatology measured with the PHQ-9 questionnaire | 12 months
  9 questions corresponding to the Diagnostic Statistical Manual symptoms for major depressive disorder during the past 2 weeks. The PHQ-9 score can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day).
Health related quality of life with the EuroQol 5-Dimension 5-Level questionnaire | 12 months
  EQ-5D-5L: covers the dimensions mobility, self-care, daily activities, pain and discomfort, and anxiety and depression. It contains a five response level: "no problems" to "not able to". Scores will be converted to a single utility index score using the value set of the Netherlands to obtain scores on a formative scale from 0 (lowest quality of life) to 1 (highest quality of life). The visual analog scale (VAS) is included for marking overall health today.
Wellbeing with the ICEpop CAPability questionnaire | 12 months
  ICECAP-O: it measures five capability dimensions: attachment, security, role, enjoyment, and control. With one question per dimension. Each dimension can be scored on four levels. An overall score can range from 0 to 1, with higher scores indicating better capability.
Health literacy with the European Health Literacy Survey Questionnaire | 12 months
  HLS-EU-Q: 16 items, they can be scored from "very easy" to "very difficult". Scoring varies between 0 and 16. Higher scores meaning more difficulty.

OTHER OUTCOMES:
Health care utilization with the Medical Cost Questionnaire | 12 months
  The iMCQ is an instrument for measuring medical consumption. The iMCQ includes 35 questions on how often patients have contact with health care providers over the last 3 months.
Process evaluation: questionnaire based on both the RE-AIM framework and Telemonitoring Acceptance Framework | 6 months
  For the intervention group, a process evaluation will take place by using a questionnaire with 22 questions, which is developed based on both the RE-AIM framework and Telemonitoring Acceptance Framework. Three essential features of understanding the process through which outcomes are achieved will be identified: 1) context, 2) implementation and 3) mechanisms of impact. In addition, elements from the Telemonitoring Acceptance Framework will be used to assess trust, behavioral intention, self-efficacy, performance expectancy, effort expectancy, social influence, facilitating conditions, technology anxiety, hedonic motivation and user opinions regarding the nurse-assisted online eye-screening tool.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth van Nispen, Principal Investigator — Amsterdam UMC - VUmc
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

REFERENCES:
- [Derived] Rooth V, van der Aa H, Wisse RPL, Maarsingh OR, Koopmanschap M, Keunen JEE, Vermeulen H, Klaver CCW, Janssen G, van Rens GHMB, van Nispen RMA. Health economic evaluation of a nurse-assisted online eye screening in home healthcare to reduce avoidable vision impairment (iScreen): study protocol for a cluster randomized controlled trial. Trials. 2024 Feb 2;25(1):102. doi: 10.1186/s13063-023-07882-0. PMID 38308377